CLINICAL TRIAL: NCT03083691
Title: A Phase II Trial of Nivolumab in Combination With Ipilimumab to Evaluate Efficacy and Safety Relapsed in Lung Cancer and to Evaluate Biomarkers Predictive for Response to Immune Checkpoint Inhibition
Brief Title: BIOLUMA: Biomarkers for Nivolumab and Ipilimumab and Evaluation of the Combination in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lung Cancer Group Cologne (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-2785; 2016-003334-25 (EudraCT Number)
Record Dates: First submitted 2017-03-02; First posted 2017-03-20 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell Lung
Keywords: Nivolumab; Ipilimumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: The treatment period is subdivided in Treatment Part A and B which differ between the two cohorts:
  Cohort 1 (non-squamous NSCLC):
  During Treatment Part A nivolumab 240 mg IV q2w as monotherapy is administered. At time of disease progression another re-biopsy is mandatory before initiation of combination therapy (Treatment Part B). Within Treatment Part B, nivolumab is given in a dose of 3 mg/kg q2w together with ipilimumab 1 mg/kg IV q6w.
  Cohort 2 (SCLC):
  Patients have to undergo a prescreening for high Tumor Mutation Burden. Within Treatment Part A, nivolumab 1 mg/kg q3w together with ipilimumab 3 mg/kg q3w for a total of four doses is administered. After the four combined doses have been administered, another re-biopsy is mandatory before initiation of Treatment Part B. In Treatment Part B, nivolumab 240 mg q2w monotherapy is administered until disease progression or unacceptable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1, NSCLC (Other): During Treatment Part A nivolumab 240 mg IV q2w as monotherapy is administered. At the time of disease progression a re-biopsy is performed before initiation of combination therapy (Treatment Part B). Within Treatment Part B, nivolumab is given in a dose of 3 mg/kg q2w together with ipilimumab 1 mg/kg IV q6w.
  Interventions: Drug: Nivolumab, Ipilimumab
- Cohort 2, SCLC (Other): Within Treatment Part A, nivolumab 1 mg/kg q3w together with ipilimumab 3 mg/kg q3w for a total of four doses is administered. After the four combined doses have been administered, a re-biopsy is performed before initiation of Treatment Part B. In Treatment Part B, nivolumab 240 mg q2w monotherapy is administered until disease progression or unacceptable toxicity
  Interventions: Drug: Nivolumab, Ipilimumab

INTERVENTIONS:
Drug: Nivolumab, Ipilimumab — Cohort 1: addition of ipilimumab in case of progression on nivolumab monotherapy.
  Arms: Cohort 1, NSCLC
Drug: Nivolumab, Ipilimumab — Cohort 2: upfront combination therapy of nivolumab and ipilimumab for four cycles, followed by nivolumab monotherapy.
  Arms: Cohort 2, SCLC

SUMMARY:
BIOLUMA is a multicentric non-randomised phase II trial in patients with non-squamous non-small cell lung cancer (NSCLC) (Cohort 1) and patients with small-cell lung cancer (SCLC) (Cohort 2) after failure of platinum-based first-line therapy. NSCLC patients are treated with nivolumab until disease progression and subsequently receive a combination therapy of nivolumab and ipilimumab. SCLC patients receive four cycles of nivolumab in combination with ipilimumab and subsequent nivolumab monotherapy. Primary endpoint for both cohorts is overall response rate of combination therapy.

Within the diagnostic part tumor biopsies will be analysed. Tumor tissue will be obtained before initiation of therapy and after progression on nivolumab monotherapy before addition of ipilimumab in Cohort 1 and after completion of the four nivolumab/ipilimumab combination cycles before continuation of nivolumab monotherapy in Cohort 2, respectively. Flow cytometry of blood samples and microbiome analysis of deep rectal swaps are performed prior to therapy as well as during course of treatment.

Cohort 1 (NSCLC) is closed for enrollment due to Sponsor decision.

In Cohort 2 (SCLC) a prescreening for high Tumor Mutation Burden is necessary before enrollment.

DETAILED DESCRIPTION:
Cohort 2 (SCLC) has been subdivided by amendment in Cohort 2a without prescreening and Cohort 2b with TMB-prescreening. For Cohort 2a enrollment has been stopped in December 2017. Cohort 2b is closed for enrollment as the cohort is fully recruited.

ELIGIBILITY:
Note: Both cohorts are closed for enrollment

Inclusion Criteria:

* Cohort 1: Subjects with histologically or cytologically confirmed advanced non-squamous non-small cell lung cancer who present with stage IIIB or stage IV disease after failure of platinum-based first-line therapy. Subjects who received adjuvant/neoadjuvant therapy or definitive chemoradiation and develop recurrence or progression, with evidence of stage IIIB-IV disease within 6 months after completion of therapy, are eligible.
* Cohort 2: Subjects in Cohort 2 have to undergo Prescreening to determine Tumor Mutation Burden. Only patients with high Tumor Mutation Burden are eligible.

Subjects with histologically or cytologically confirmed limited-stage or extensive-stage small cell lung cancer after failure of platinum-based first-line therapy.

Cohort 1 and Cohort 2:

* Signed and dated written informed consent form must be obtained before the performance of any study-specific procedure
* Male or female patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Subjects must be willing to undergo the baseline biopsie during screening, if medically feasible
* Measurable disease by CT or MRI per RECIST 1.1 criteria.
* Screening laboratory values must meet the following criteria and should be obtained within 28 days prior to registration: white blood cell count ≥ 2000/μL, Neutrophils ≥ 1500/μL, Platelets ≥ 100 x103/μL, Hemoglobin > 9.0 g/dL, Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min, AST/ALT ≤ 3 x ULN for patients without liver metastasis, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 x ULN for patients with liver metastasis, Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Prior chemotherapy must have been completed at least 4 weeks before study drug administration, and all AEs have either returned to baseline or stabilized.
* Prior palliative radiotherapy must have been completed at least 14 days prior to study drug administration
* Prior targeted therapy must have been completed at least 4 weeks prior to study drug administration
* Cohort 1 and 2a: Subjects with central nervous system (CNS) metastasis are eligible if CNS metastases are treated and subjects have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 28 days prior to first dose of study drug administration. In addition, subjects must either be off corticosteroids or on a stable dose or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).

Cohort 2b: Subjects with CNS metastases are eligible. Radiation of CNS metastases at initiation of study drug treatment is allowed if the trial subject has target lesions outside of the brain.

* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception and must agree to use adequate method to avoid pregnancy for 5 month after the last dose of study drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of b-HCG) within 24 hours prior to the start of nivolumab.
* Women must not be breastfeeding.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP must be willing to adhere to contraception for a period of 7 month post treatment completion.

Exclusion Criteria:

* Subjects with squamous cell NSCLC
* Cohort 1: activating epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) translocation
* Cohort 1 and 2a only: More than one prior line of chemotherapy for treatment of advanced disease Note for Cohort 2b: inclusion of patients who received 2nd line treatment is allowed if 2nd line did not include an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA-4 antibody as monotherapy or in combination with other than platinum-based chemotherapy.
* Medical conditions associated with significantly increased risk for bleeding complications caused by biopsy procedures (e.g. known coagulopathies, therapeutic anticoagulation)
* Cohort 1 and 2a only: Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for 4 weeks after treatment is complete and within 28 days prior to the first dose of study drug administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Presence or history of any other primary malignancy other than NSCLC for Cohort 1 and SCLC for Cohort 2 within 5 years prior to enrolment into the trial, except for adequately treated basal or squamous cell carcinoma of the skin or any adequately treated in situ carcinoma.
* Active, known or suspected autoimmune disease. Subjects are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Positive test for hepatitis B or hepatitis C indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.

Note for Cohort 2b: higher doses of corticosteroids for patients receiving radiation therapy of brain metastases are allowed.

* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.

Note: SCLC-Patients who where treated with a combination therapy of platinum-based chemotherapy together with anti-PD-1/PD-L1 treatment are eligible.

* Prisoners or subjects who are involuntarily incarcerated.
* Any other serious or uncontrolled medical disorder, active infections, physical exam findings, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability or study results.
* Allergies and Adverse Drug Reaction: History of allergy to study drug components and history of severe hypersensitivity reaction to any monoclonal antibody
* Current treatment within another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Cohort 1: ORR after addition of ipilimumab to nivolumab treatment. | From beginning of combination therapy until the date of first documented progression, or date of death of any cause, whichever occurs first, assessed up to 120 months.
  ORR is defined as proportion of patients with reduction in tumor burden as assessed by RECIST 1.1 criteria (investigator-assessed).
Cohort 2: ORR of the combination therapy nivolumab and ipilimumab. | From beginning of combination therapy until the date of first documented progression, or date of death of any cause, whichever occurs first, assessed up to 120 months.
  ORR is defined as proportion of patients with reduction in tumor burden as assessed by RECIST 1.1 criteria (investigator-assessed).

SECONDARY OUTCOMES:
Overall survival of nivolumab monotherapy/nivolumab + ipilimumab combination therapy | From date of first dose until death, withdrawal of informed consent or lost to follow-up, through study completion, an average of 1 year, up to 120 months.
  Time from date of first dose to the date of death to any cause.
Progression-free survival of nivolumab monotherapy/nivolumab + ipilimumab combination therapy | From date of first dose to first documentation of objective disease progression or to death on study due to any cause, an average of 6 months, up to 120 months.
  Time from the date of first dose to first documentation of objective disease progression or to death on study due to any cause, whichever occurs first.
Duration of response of nivolumab monotherapy/nivolumab + ipilimumab combination therapy | First on-study tumor assessment is performed at Week 9 in Cohort 1 and at Week 5 in Cohort 2 and subsequently every 8 weeks through study completion, an average of 1 year.
  Time from the first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the first documentation of objective disease progression or to death due to any cause, whichever occurs first
Incidence, severity and grading of adverse events (AEs) during nivolumab monotherapy/ nivolumab + ipilimumab combination therapy | From initiation of study drug, continuously during the treatment period and for a minimum of 100 days following the last dose of study treatment.
  Adverse events are documented according to the Common Terminology Criteria for Adverse Events (CTCAE)
Incidence, severity and grading of serious adverse events (SAEs) during nivolumab monotherapy/ nivolumab + ipilimumab combination therapy | Following the subject's written consent, SAEs are collected that occur within survival follow-up through study completion, an average of 6 months. For subjects who did not receive study medication, SAEs are collected until resolved.
  Serious adverse events are documented according to the Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wolf, MD, Principal Investigator — University ClinicCologne
Locations (16):
- Germany (16):
  - SLK-Fachklinik Löwenstein, Löwenstein, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Innere Medizin VIII - Medizinische Onkologie und Pneumologie, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Würzburg - Comprehensive Cancer Center Mainfranken, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt - Medizinische Klinik II, Frankfurt am Main, Hesse
  - Klinikum Kassel - Klinik für Hämatologie und Onkologie, Kassel, Hesse
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Uniklinik RWTH - Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzellentransplantation, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Bonn - Medizinische Klinik und Poliklinik III, Bonn, North Rhine-Westphalia
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln - Lungenkrebszentrum Köln-Merheim, Cologne, North Rhine-Westphalia
  - St.-Johannes-Hospital Dortmund, Dortmund, North Rhine-Westphalia
  - Uniklinik Düsseldorf - Klinik für Hämatologie und Onkologie, Düsseldorf, North Rhine-Westphalia
  - Lungenklinik Hemer, Hemer, North Rhine-Westphalia
  - Universitätsklinikum Münster - Medizinische Klinik A, Pneumologie, Münster, North Rhine-Westphalia
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg, Schleswig-Holstein
  - Evangelische Lungenklinik Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No